CLINICAL TRIAL: NCT02670551
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter, Fixed-Dose Clinical Trial Evaluating The Efficacy, Safety And Tolerability Of Cariprazine In Patients With Bipolar I Depression
Brief Title: Study on the Efficacy, Safety, and Tolerability of Cariprazine Relative to Placebo in Participants With Bipolar I Depression
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RGH-MD-54; 2016-000757-13 (EudraCT Number)
Record Dates: First submitted 2016-01-28; First posted 2016-02-01 (Estimated); Results first posted 2019-01-30 (Actual); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Bipolar Disorder; Depression
MeSH Terms: conditions — Bipolar Disorder; Depression | interventions — cariprazine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Placebo (Placebo Comparator): Following a 7 to 14 days screening/washout period, placebo-matching cariprazine capsule, one per day, orally for 6 weeks.
  Interventions: Drug: Placebo
- Cariprazine 1.5 mg (Experimental): Following a 7 to 14 days screening/washout period, cariprazine 1.5 milligram (mg) capsule, one per day, orally for 6 weeks.
  Interventions: Drug: Cariprazine
- Cariprazine 3.0 mg (Experimental): Following a 7 to 14 days screening/washout period, cariprazine 1.5 mg capsule, one per day for 2 weeks followed by cariprazine 3.0 milligram (mg) capsule, one per day, orally beginning on Day 15 for 4 weeks.
  Interventions: Drug: Cariprazine

INTERVENTIONS:
Drug: Cariprazine
  Other Names: VRAYLAR®
  Arms: Cariprazine 1.5 mg; Cariprazine 3.0 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
This study investigates the efficacy of a fixed-dose regimen of cariprazine 1.5 milligram (mg)/day or 3 mg/day compared to placebo for treatment of the depressive episode in participants with bipolar I disorder. The safety and tolerability of the fixed-dose regimens will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Currently meet the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) criteria for bipolar I disorder without psychotic features confirmed by the administration of the Mini International Neuropsychiatric Interview (MINI), with a current major depressive episode of at least 4 weeks and not exceeding 12 months in duration
* Currently treated as an outpatient at the time of enrollment
* A verified previous manic or mixed episode. Verification must include one of the following sources: --Treatment of mania with an anti-manic agent (eg, lithium or divalproate) or antipsychotic medication with an approved indication for mania --Hospital records/Medical records --Participant report corroborated by caretaker or previous or current treating clinician
* 17-item Hamilton Depression Rating Scale (HAMD-17) total score ≥ 20
* HAMD-17 item 1 score ≥ 2
* Clinical Global Impressions-Severity (CGI-S) score ≥ 4
* Negative serum β-human chorionic gonadotropin (β-hCG) pregnancy test (women of childbearing potential only)
* Normal physical examination, clinical laboratory test results, and electrocardiogram (ECG) results or abnormal findings that are judged not clinically significant by the Principal Investigator (PI)

Exclusion Criteria:

* Young Mania Rating Scale (YMRS) total score > 12
* Four or more episodes of a mood disturbance (depression, mania, hypomania, or mixed state) within the 12 months before Visit 1
* Any current axis 1 psychiatric diagnosis other than bipolar disorder with the exception of specific phobias
* History of meeting DSM-5 criteria for: ○ Dementia, amnesic, or other cognitive disorder ○ Schizophrenia, schizoaffective, or other psychotic disorder

  ○ Mental retardation - DSM-5-based diagnosis of borderline or antisocial personality disorder or other axis II disorder of sufficient severity to interfere with participation in this study
* History of meeting DSM-5 criteria for alcohol or substance abuse or dependence (other than nicotine or caffeine) within the 6 months before Visit 1
* Positive result on blood alcohol test or urine drug screen for any prohibited medication. Exception: ○ Participants with a positive cannabinoid on entry may be retested before randomization. If the participant remains positive, the participant is no longer eligible ○ Participants positive for opiates on entry, discussion with Study Physician is required.
* Electroconvulsive therapy in the 3 months before Visit 1
* Previous lack of response to electroconvulsive therapy
* Treatment with a depot antipsychotic drug within 1 treatment cycle before Visit 1
* Treatment with clozapine in a dose of > 50 mg/day in the past 2 years
* Prior participation in any investigational study of RGH-188 or cariprazine within the past 12 months
* Previous treatment with vagus nerve stimulation or transcranial magnetic stimulation within 6 months before Visit 1
* Prior participation with any clinical trials, involving experimental or investigational drugs, within 6 months before Visit 1 or during the study
* Initiation or termination of psychotherapy for depression within the 3 months preceding Visit 1, or plans to initiate, terminate, or change such therapy during the course of the study.
* Pregnant, breastfeeding, or planning to become pregnant or breastfeed during the study
* Gastric bypass or any condition that would be expected to affect drug absorption (lap band procedures are acceptable if there is no problem with absorption)
* Known history of cataracts or retinal detachment
* Known human immunodeficiency virus infection
* Employee, or immediate relative of an employee, of the Sponsor, any of its affiliates or partners, or the study center

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2016-03-17 (Actual); Primary Completion 2017-07-19 (Actual); Study Completion 2017-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clincial Director, Study Director — Forest Research Institute, Inc., an affiliate of Allergan, plc
Locations (74):
- United States (44):
  - Arkansas Psychiatric Clinic Clinical Research Trials PA, Little Rock, Arkansas
  - ATP Clinical Research, Inc., Costa Mesa, California
  - Synergy San Diego, Escondido, California
  - Integrated Medical and Behavioral Associates, Glendale, California
  - Apostle Clinical Trials, Inc., Long Beach, California
  - Pacific Research Partners, LLC, Oakland, California
  - Artemis Institute for Clinical Research, San Diego, California
  - Schuster Medical Research Institute, Sherman Oaks, California
  - Viking Clinical Research, Temecula, California
  - Pacific Clinical Research Medical Group, Upland, California
  - Comprehensive Psychiatric Care, Norwich, Connecticut
  - CNS Healthcare, Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - Olympian Clinical Research, Tampa, Florida
  - Radiant Research, Atlanta, Georgia
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Northwest Behavioral Research Center, Marietta, Georgia
  - Carman Research, Smyrna, Georgia
  - Psychiatric Medicine Associates, L.L.C, Skokie, Illinois
  - Neuroscience Research Institute Inc., Winfield, Illinois
  - St. Charles Psychiatric Associates - Midwest Research Group, Saint Charles, Missouri
  - Altea Research Institute, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - Neurobehavioral Research, Inc., Cedarhurst, New York
  - Medical & Behavioral Health Research, PC, New York, New York
  - Neuro-Behavioral Clinical Research, Canton, Ohio
  - Patient Priority Clinical Sites, Cincinnati, Ohio
  - Ohio State University Department of Psychiatry, Columbus, Ohio
  - Midwest Clinical Research Center, Dayton, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Oregon Center for Clinical Investigations, Inc., Portland, Oregon
  - Oregon Center for Clinical Investigations, Salem, Oregon
  - Lehigh Center for Clinical Research, Allentown, Pennsylvania
  - Lincoln Research, LLC, Lincoln, Rhode Island
  - Clinical Neuroscience Solutions, Memphis, Tennessee
  - Red Oak Psychiatry Associates, PA, Houston, Texas
  - Houston Clinical Trials, LLC, Houston, Texas
  - Research Across America, Plano, Texas
  - Family Psychiatry of The Woodlands, The Woodlands, Texas
  - Alliance Research Group, Richmond, Virginia
  - Northwest Clinical Research Center, Bellevue, Washington
  - Core Clinical Research, Kirkland, Washington
  - Summit Research Network Seattle, Seattle, Washington
- Bulgaria (13):
  - Mental Health Centre 'Prof. Dr. Ivan Temkov', EOOD, Burgas
  - SPH - Kardzhali, EOOD, Kardzhali
  - MHAT "Dr. Hristo Stambolski", EOOD, Kazanlak
  - State Psychiatric Hospital - Lovech, Lovech
  - UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - UMHAT "Sv. Georgi", EAD, Plovdiv
  - MHC - Ruse, EOOD, Rousse
  - MHATNP "Sv.Naum", EAD, Sofia
  - UMHAT "Alexandrovska" EAD, Sofia
  - Military Medical Academy - MHAT - Sofia, Sofia
  - Medical Centre "Doverie" AD, Sofia
  - MHAT-Targovishte, AD, Targovishte
  - DCC "Mladost M" - Varna, OOD, Varna
- Estonia (3):
  - Marienthal Center of Psychiatry and Psychology, Tallinn
  - West Tallinn Central Hospital, Tallinn
  - Tartu University Hospital, Tartu
- Lithuania (5):
  - Romuvos klinika, UAB, Kaunas
  - Neuromeda, JSC, Kaunas
  - Republican Kaunas Hospital Psychiatry Clinic Mariu Division, Public Institution, Kaunas
  - Hospital of Lithuanian University of Health Sciences Kaunas Clinics, Kaunas
  - 232Antakalnis Psychiatric Consultation Center, Public Institution, Vilnius
- Poland (8):
  - Podlaskie Centrum Psychogeriatrii, Bialystok
  - Przychodnia Srodmiescie Sp. z o. o., Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Niepubliczny Zaklad Opieki Psychiatrycznej MENTIS, Leszno
  - Clinical Best Solutions, Lublin
  - Specjalistyczna Praktyka Lekarska Marek Domański, Lublin
  - NZOZ Syntonia, Pruszcz Gdański
  - Torunskie Centrum Psychiatrii Neuromed, Torun
- INSPIRA Clinical Research, San Juan, Puerto Rico

REFERENCES:
- [Derived] McIntyre RS, Llorca PM, Aronin LC, Yu J, Nguyen HB. Effect of Cariprazine on Anhedonia in Patients with Bipolar I Depression: Post Hoc Analysis of Three Randomized Placebo-Controlled Clinical Trials. Adv Ther. 2025 Jan;42(1):246-260. doi: 10.1007/s12325-024-03009-2. Epub 2024 Nov 9. PMID 39520655
- [Derived] Citrome L, Yatham LN, Patel MD, Barabassy A, Hankinson A, Earley WR. Cariprazine and akathisia, restlessness, and extrapyramidal symptoms in patients with bipolar depression. J Affect Disord. 2021 Jun 1;288:191-198. doi: 10.1016/j.jad.2021.03.076. Epub 2021 Mar 31. PMID 33915374
- [Derived] Thase ME, Harrington A, Calabrese J, Montgomery S, Niu X, Patel MD. Evaluation of MADRS severity thresholds in patients with bipolar depression. J Affect Disord. 2021 May 1;286:58-63. doi: 10.1016/j.jad.2021.02.043. Epub 2021 Feb 20. PMID 33677183
- [Derived] Yatham LN, Vieta E, McIntyre RS, Jain R, Patel M, Earley W. Broad Efficacy of Cariprazine on Depressive Symptoms in Bipolar Disorder and the Clinical Implications. Prim Care Companion CNS Disord. 2020 Sep 17;22(5):20m02611. doi: 10.4088/PCC.20m02611. PMID 32942346
- [Derived] Earley WR, Burgess M, Rekeda L, Hankinson A, McIntyre RS, Suppes T, Calabrese JR, Yatham LN. A pooled post hoc analysis evaluating the safety and tolerability of cariprazine in bipolar depression. J Affect Disord. 2020 Feb 15;263:386-395. doi: 10.1016/j.jad.2019.11.098. Epub 2019 Nov 22. PMID 31969269
- [Derived] Earley W, Burgess MV, Rekeda L, Dickinson R, Szatmari B, Nemeth G, McIntyre RS, Sachs GS, Yatham LN. Cariprazine Treatment of Bipolar Depression: A Randomized Double-Blind Placebo-Controlled Phase 3 Study. Am J Psychiatry. 2019 Jun 1;176(6):439-448. doi: 10.1176/appi.ajp.2018.18070824. Epub 2019 Mar 8. PMID 30845817

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Total 782 participants were screened for eligibility; 488 participants randomized to receive double-blind treatment; 480 participants received at least 1 dose of double-blind treatment (Safety Population) and 474 participants had at least 1 postbaseline Montgomery-Åsberg Depression Rating Scale total score assessment (Intent-to-Treat Population).
Groups:
- Cariprazine 3.0 mg: Following a 7 to 14 days screening/washout period, cariprazine 1.5 mg capsule, one per day for 2 weeks followed by cariprazine 3.0 mg capsule, one per day, orally beginning on Day 15 for 4 weeks.
Period: Overall Study
Arm/Group | Placebo | Cariprazine 1.5 mg | Cariprazine 3.0 mg
Started | 163 | 160 | 165
Received Treatment (Safety Population) | 158 | 157 | 165
Completed | 135 | 134 | 134
Not Completed | 28 | 26 | 31
Not completed — Adverse Event | 4 | 7 | 9
Not completed — Lack of Efficacy | 2 | 0 | 3
Not completed — Withdrawal of Consent | 6 | 3 | 8
Not completed — Lost to Follow-up | 5 | 7 | 6
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Noncompliance with study drug | 3 | 3 | 2
Not completed — Other Miscellaneous Reasons | 2 | 3 | 3
Not completed — Did Not Receive Treatment | 5 | 3 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants who were randomized to receive the double-blind treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Cariprazine 1.5 mg | Cariprazine 3.0 mg | Total
Number analyzed (Participants) | 163 | 160 | 165 | 488
Age, Continuous [Mean (Full Range); unit: years] | 43.9 [18 to 65] | 42.6 [18 to 65] | 41.9 [19 to 64] | 42.8 [18 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 101 | 94 | 289
  Male | 69 | 59 | 71 | 199
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 118 | 126 | 126 | 370
  Black or African American | 39 | 29 | 37 | 105
  Asian | 3 | 2 | 0 | 5
  American Indian or Alaska Native | 1 | 1 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 0 | 2
  Multiple | 0 | 2 | 1 | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 15 | 14 | 42
  Not Hispanic or Latino | 150 | 145 | 151 | 446
Montgomery-Åsberg Depression Rating Scale (MADRS) Score at Baseline [Mean (Standard Deviation); unit: score on a scale] — The Montgomery-Åsberg Depression Rating Scale is a 10-item, clinician-rated scale that evaluates the participant's depressive symptomatology during the past week. Participants were rated on items assessing feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty in concentration, and lack of interest. Each of the 10 items was scored on a 7-point scale with a score of 0 reflecting no symptoms and a score of 6 reflecting symptoms of maximum severity for a total possible score of 0 (best) to 60 (worst). Population: Montgomery-Åsberg Depression Rating Scale (MADRS) score at Baseline was analyzed for ITT population.
  score on a scale
    number analyzed (Participants) | 156 | 154 | 164 | 474
    (all) | 30.3 (4.5) | 30.6 (4.2) | 31.1 (4.8) | 30.7 (4.5)
Clinical Global Impressions-Severity (CGI-S) Score at Baseline [Mean (Standard Deviation); unit: score on a scale] — The Clinical Global Impressions-Severity (CGI-S) is a clinician-rated scale that measures the overall severity of a participant's illness in comparison with the severity of other participants the physician has observed. The participant was rated on a scale from 1 to 7, with 1 indicating a "normal state" and 7 indicating "among the most extremely ill participants." Population: Clinical Global Impressions-Severity (CGI-S) score at Baseline was analyzed for ITT population.
  score on a scale
    number analyzed (Participants) | 156 | 154 | 164 | 474
    (all) | 4.5 (0.5) | 4.5 (0.5) | 4.5 (0.5) | 4.5 (0.5)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Montgomery-Åsberg Depression Rating Scale (MADRS) Score at Week 6
Description: The Montgomery-Åsberg Depression Rating Scale (MADRS) is a 10-item, clinician-rated scale that evaluates the participant's depressive symptomatology during the past week. Participants were rated on items assessing feelings of sadness, lassitude, pessimism, inner tension, suicidality, reduced sleep or appetite, difficulty in concentration, and lack of interest. Each of the 10 items was scored on a 7-point scale with a score of 0 reflecting no symptoms and a score of 6 reflecting symptoms of maximum severity for a total possible score of 0 (best) to 60 (worst). A negative change from Baseline indicates improvement.
Time Frame: Baseline (Week 0) to Week 6
Population: The Intent-to-Treat (ITT) Population included all participants from the safety population who had at least 1 postbaseline assessment of the MADRS total score. Overall number of participants analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Cariprazine 1.5 mg | Cariprazine 3.0 mg
Number analyzed (Participants) | 137 | 135 | 136
score on a scale | -12.6 (0.76) | -15.1 (0.77) | -15.6 (0.76)
Statistical Analysis 1: Comparison: Placebo vs Cariprazine 1.5 mg; To control the overall type I error rate for multiple comparisons of 2 active doses versus placebo at Week 6 for the primary and secondary efficacy parameters, the parallel gatekeeping procedure was implemented; Test type: Superiority; p = 0.0331, Mixed Model Repeated Measures (MMRM) — MMRM analysis was used. Fixed factors: treatment group, pooled study center, visit, treatment-group-by-visit interaction. Covariates: Baseline value, baseline value-by-visit interaction. P-value was adjusted by matched parallel gatekeeping procedure; Least Squares Mean Difference = -2.5, 95% CI 2-sided [-4.6 to -0.4]
Statistical Analysis 2: Comparison: Placebo vs Cariprazine 3.0 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0103, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -3.0, 95% CI 2-sided [-5.1 to -0.9]

2. Secondary Outcome: Change From Baseline in Clinical Global Impressions-Severity (CGI-S) Score at Week 6
Description: The Clinical Global Impressions-Severity (CGI-S) is a clinician-rated scale that measures the overall severity of a participant's illness in comparison with the severity of other participants the physician has observed. The participant was rated on a scale from 1 to 7, with 1 indicating a "normal state" and 7 indicating "among the most extremely ill participants." A negative change from Baseline indicates improvement.
Time Frame: Baseline (Week 0) to Week 6
Population: ITT Population included all participants from the safety population who had at least 1 postbaseline assessment of the MADRS total score. Overall number of participants analyzed is the number of participants with data available for analysis at the given time-point.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | Cariprazine 1.5 mg | Cariprazine 3.0 mg
Number analyzed (Participants) | 137 | 135 | 136
score on a scale | -1.3 (0.09) | -1.6 (0.10) | -1.6 (0.09)
Statistical Analysis 1: Comparison: Placebo vs Cariprazine 1.5 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0714, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.2, 95% CI 2-sided [-0.5 to 0.0]
Statistical Analysis 2: Comparison: Placebo vs Cariprazine 3.0 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0662, Mixed Model Repeated Measures (MMRM) — [p-value comment as in outcome 1, analysis 1]; Least Squares Mean Difference = -0.3, 95% CI 2-sided [-0.5 to -0.0]

ADVERSE EVENTS:
Time Frame: First dose to 30 days past last dose (Up to 80 Days)
Description: Safety Population included all participants in the randomized population who took at least 1 dose of double-blind investigational product.
Arm/Group | Placebo | Cariprazine 1.5 mg | Cariprazine 3.0 mg
All-Cause Mortality (participants affected / at risk) | 0/158 | 0/157 | 0/165
Serious Adverse Events (participants affected / at risk) | 2/158 | 2/157 | 2/165
Other Adverse Events (participants affected / at risk) | 43/158 | 48/157 | 62/165
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=158) | Cariprazine 1.5 mg (N=157) | Cariprazine 3.0 mg (N=165)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Chronic tonsillitis (Infections and infestations) | 1 | 0 | 0
Bipolar disorder (Psychiatric disorders) | 0 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=158) | Cariprazine 1.5 mg (N=157) | Cariprazine 3.0 mg (N=165)
Nausea (Gastrointestinal disorders) | 1 | 6 | 15
Dry mouth (Gastrointestinal disorders) | 9 | 6 | 3
Headache (Nervous system disorders) | 13 | 7 | 12
Akathisia (Nervous system disorders) | 5 | 10 | 9
Dizziness (Nervous system disorders) | 3 | 8 | 6
Somnolence (Nervous system disorders) | 3 | 8 | 6
Sedation (Nervous system disorders) | 2 | 8 | 5
Insomnia (Psychiatric disorders) | 11 | 7 | 12
Restlessness (Psychiatric disorders) | 6 | 2 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.

DOCUMENTS (2):
  • Study Protocol (2016-02-17): https://cdn.clinicaltrials.gov/large-docs/51/NCT02670551/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-29): https://cdn.clinicaltrials.gov/large-docs/51/NCT02670551/SAP_001.pdf